CLINICAL TRIAL: NCT06412380
Title: Influence of High Insertion Torque and Type of Bone on Post-operative Pain and Survival Rate of Dental Implants
Brief Title: Influence of Insertion Torque and Bone Type on Post-operative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sharjah (Other)
Collaborators: Yarmouk University (Other)
Responsible Party: Principal Investigator, Ahmed Aziz, Assistant Professor, University of Sharjah
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 210
Record Dates: First submitted 2024-05-08; First posted 2024-05-14 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Postoperative Pain; Postsurgical Pain; Dental Implant Failed
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain level (Experimental): After implant placement, all participants were requested to record their pain level using the 10-cm visual analog scale (VAS) ranging from 0 "no pain" to 10 "worst pain ever." The scale had no other markings along the line. Patients were asked to record their pain level after surgery, 24 hours after surgery, at day 2, day 4 and at week 1, week 2, and week 3.
  Interventions: Procedure: Implant insertion
- Implant torque (Experimental): Implants were classified into 4 groups based on the IT value; Low: 58 implants (10-29 Ncm); Regular: 95 implants (30-50 Ncm); High: 46 implants (51-100 Ncm); and Very High: 31 implants (101-180 Ncm).
  Interventions: Procedure: Implant insertion

INTERVENTIONS:
Procedure: Implant insertion — All patients received a single Tapered Screw implant (Bioinnovation Dental®, Brazil). The implants were placed according to the manufacturer's instructions by using the appropriate burs with a final master drill of 3.5 or 4.5 mm in diameter by one senior oral surgeon. These implants were multi-threaded, and their surfaces were both sandblasted and acid etched. Of the 230 participants, 172 received a single 5 x 10-mm implant, and 58 received a 4 x 10-mm implant.
  Other Names: Implant surgery

SUMMARY:
The objectives of this clinical study were to assess the effect of different ITs and bone types on POP levels and survival rates and to investigate the effect of different patient- and site-related factors on POP levels and survival rates.

DETAILED DESCRIPTION:
This prospective clinical study included 230 patients treated with a single tapered screw implant (Bioinnovation Dental®, Brazil). The implants were placed using the appropriate burs with a final master drill of 3.5 or 4.5 mm in diameter by one senior oral surgeon. These implants were multi-threaded, and their surfaces were both sandblasted and acid etched. Of the 230 participants, 172 received a single 5 x 10-mm implant, and 58 received a 4 x 10-mm implant.

For the higher torque range (90 - 200 Ncm), the maximum IT was recorded with an electronic digital torque measuring device (Tohnichi BTGE200CN-G, Hitachi, Japan), while a different gauge (Tohnichi BTG90CN-S, Hitachi, Japan) was used for the lower torque range (10 - 90 Ncm). All implants were placed at the crestal level and closed with a cover screw, and the flap was then sutured with non-resorbable 4/0 nylon suture (Resorba® Germany).

Pain levels were recorded at day 1, 2 and 4 and at week 1, 2 and 3 after surgery using visual analog scale (VAS) ranging from 0 "no pain" to 10 "worst pain ever. Implants were classified into 4 groups based on the IT value; Low: 60 implants (10-29 Ncm, mean=15 Ncm); Regular: 102 implants (30-50 Ncm, mean=42 Ncm); High: 47 implants (51-100 Ncm, mean=75 Ncm); and Very high: 21 implants (101-200 Ncm, mean=170 Ncm).

Implant survival was assessed clinically and radiographically at 3, 6, 12, 24 and 36 months. The criteria for implant success according to Buser et al, were no radiolucent zone around the implant, confirmed individual implant stability, and no suppuration, pain or ongoing pathologic processes. All implants that failed to fulfill these success criteria were regarded as failures.

The effect of IT, bone type, implant location, age, gender and smoking was measured with regression analysis. Kaplan-Meier survival analysis was performed to calculate the overall implant survival probabilities. The level of statistical significance was set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* partially edentulous patients who presented with one or more missing teeth in the maxillary or mandibular jaw
* at least18 years old, adequate oral hygiene
* absence of infection or periodontal problems adjacent to the implant site - sufficient bone thickness with a minimum 6-mm width and 12-mm length to accommodate implants of 4 or 5 mm in diameter and 10 mm in length.

Exclusion Criteria:

* uncontrolled diabetes
* hypertension
* pregnancy
* bone diseases
* use of bisphosphonates
* heavy smoker (more than 20 cigarettes /day)
* severe alcohol or drug use
* patients with recent extraction of teeth and patients requiring bone and soft tissue augmentation procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Post-operative pain | 1 month
  Pain was assessed after surgery using the 10-cm visual analog scale (VAS) ranging from 0 "no pain" to 10 "worst pain ever." The scale has no other markings along the line. Patients will be asked to record their pain level before surgery and after surgery, 24 hours after surgery, at day 2, day 4 and at week 1, week 2, and week 3.

SECONDARY OUTCOMES:
Survival rate of implants | 36 months
  Implant survival was assessed clinically and radiographically at 3, 6, 12, 24 and 36 months. The criteria for implant success according to Buser et al, were no radiolucent zone around the implant, confirmed individual implant stability, and no suppuration, pain or ongoing pathologic processes (Buser et al., 1997). All implants that failed to fulfill these criteria were regarded as failures.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Aziz, PhD, Principal Investigator — University of Sharjah
Locations (1):
- University of Sharjah, Sharjah city, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No
Individuals data will not be shared, data required normally for publication will be shared upon reasonable request.

REFERENCES:
- [Background] Al-Khabbaz AK, Griffin TJ, Al-Shammari KF. Assessment of pain associated with the surgical placement of dental implants. J Periodontol. 2007 Feb;78(2):239-46. doi: 10.1902/jop.2007.060032. PMID 17274712
- [Background] Alissa R, Sakka S, Oliver R, Horner K, Esposito M, Worthington HV, Coulthard P. Influence of ibuprofen on bone healing around dental implants: a randomised double-blind placebo-controlled clinical study. Eur J Oral Implantol. 2009 Autumn;2(3):185-99. PMID 20467629
- [Background] Augustin G, Davila S, Udilljak T, Staroveski T, Brezak D, Babic S. Temperature changes during cortical bone drilling with a newly designed step drill and an internally cooled drill. Int Orthop. 2012 Jul;36(7):1449-56. doi: 10.1007/s00264-012-1491-z. PMID 22290154
- [Background] Barewal RM, Oates TW, Meredith N, Cochran DL. Resonance frequency measurement of implant stability in vivo on implants with a sandblasted and acid-etched surface. Int J Oral Maxillofac Implants. 2003 Sep-Oct;18(5):641-51. PMID 14579951
- [Background] Barone A, Alfonsi F, Derchi G, Tonelli P, Toti P, Marchionni S, Covani U. The Effect of Insertion Torque on the Clinical Outcome of Single Implants: A Randomized Clinical Trial. Clin Implant Dent Relat Res. 2016 Jun;18(3):588-600. doi: 10.1111/cid.12337. Epub 2015 Jun 5. PMID 26043651
- [Background] Beaudette JR, Fritz PC, Sullivan PJ, Piccini A, Ward WE. Investigation of factors that influence pain experienced and the use of pain medication following periodontal surgery. J Clin Periodontol. 2018 May;45(5):578-585. doi: 10.1111/jcpe.12885. Epub 2018 Apr 16. PMID 29500837
- [Background] Becker W, Becker BE, Hujoel P, Abu Ras Z, Goldstein M, Smidt A. Prospective clinical trial evaluating a new implant system for implant survival, implant stability and radiographic bone changes. Clin Implant Dent Relat Res. 2013 Feb;15(1):15-21. doi: 10.1111/j.1708-8208.2010.00333.x. Epub 2011 Jan 11. PMID 21223489
- [Background] Berardini M, Trisi P, Sinjari B, Rutjes AW, Caputi S. The Effects of High Insertion Torque Versus Low Insertion Torque on Marginal Bone Resorption and Implant Failure Rates: A Systematic Review With Meta-Analyses. Implant Dent. 2016 Aug;25(4):532-40. doi: 10.1097/ID.0000000000000422. PMID 27129002
- [Background] Bryce G, Bomfim DI, Bassi GS. Pre- and post-operative management of dental implant placement. Part 1: management of post-operative pain. Br Dent J. 2014 Aug;217(3):123-7. doi: 10.1038/sj.bdj.2014.650. PMID 25104691
- [Background] Calandriello R, Tomatis M, Rangert B. Immediate functional loading of Branemark System implants with enhanced initial stability: a prospective 1- to 2-year clinical and radiographic study. Clin Implant Dent Relat Res. 2003;5 Suppl 1:10-20. doi: 10.1111/j.1708-8208.2003.tb00011.x. PMID 12691646